CLINICAL TRIAL: NCT00005431
Title: Coronary Heart Disease Risk Factors in Blacks Vs Whites
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4349; R03HL052204 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To use data from the Epidemiologic Follow-up Study of the National Health and Nutrition Examination Survey (NHANES) to develop models to predict morbidity and mortality as a function of risk factors for coronary artery disease. Bivariate dependent survival distributions were examined.

DETAILED DESCRIPTION:
The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-09; Study Completion 1996-02 (Actual)

REFERENCES:
- [Background] McGee D, Cooper R, Liao Y, Durazo-Arvizu R. Patterns of comorbidity and mortality risk in blacks and whites. Ann Epidemiol. 1996 Sep;6(5):381-5. doi: 10.1016/s1047-2797(96)00058-0. PMID 8915468